CLINICAL TRIAL: NCT06557785
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of CH505M5 N197D mRNA-gp160 Followed by CH505 TF mRNA-gp160 in Adults in Overall Good Health Without HIV
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of CH505M5 N197D mRNA-gp160 Followed by CH505 TF mRNA-gp160 in Adults in Overall Good Health Without HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 312; 39019 (Other: DAIDS DOCUMENT ID)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (25 mcg) (Experimental): 25 mcg of CH505M5 N197D mRNA-gp160, to be administered as a split dose intramuscularly at weeks 0, 8, and 16.
  Followed by:
  25 mcg of CH505 TF mRNA-gp160, to be administered as a split dose intramuscularly at week 24.
  Interventions: Biological: CH505M5 N197D mRNA-gp160; Biological: CH505 TF mRNA-gp160
- Group 2 (50 mcg) (Experimental): 50 mcg of CH505M5 N197D mRNA-gp160, to be administered as a split dose intramuscularly at weeks 0, 8, and 16.
  Followed by:
  50 mcg of CH505 TF mRNA-gp160, to be administered as a split dose intramuscularly at week 24.
  Interventions: Biological: CH505M5 N197D mRNA-gp160; Biological: CH505 TF mRNA-gp160
- Group 3 (100 mcg) (Experimental): 100 mcg of CH505M5 N197D mRNA-gp160, to be administered as a split dose intramuscularly at weeks 0, 8, and 16.
  Followed by:
  100 mcg of CH505 TF mRNA-gp160, to be administered as a split dose intramuscularly at week 24.
  Interventions: Biological: CH505M5 N197D mRNA-gp160; Biological: CH505 TF mRNA-gp160
- Group 4 (150 mcg) (Experimental): 150 mcg of CH505M5 N197D mRNA-gp160, to be administered as a split dose intramuscularly at weeks 0, 8, and 16.
  Followed by:
  150 mcg CH505 TF mRNA-gp160, to be administered as a split dose intramuscularly at week 24.
  Interventions: Biological: CH505M5 N197D mRNA-gp160; Biological: CH505 TF mRNA-gp160

INTERVENTIONS:
Biological: CH505M5 N197D mRNA-gp160 — To be administered intramuscularly as a split dose
Biological: CH505 TF mRNA-gp160 — To be administered intramuscularly as a split dose

SUMMARY:
This is a multicenter, open-label, non-randomized, dose escalation, first-in-human (FIH) trial to evaluate the safety and immunogenicity of CH505M5 N197D mRNA-gp160 and CH505 TF mRNA-gp160. Both products are mRNA encapsulated in lipid nanoparticles (LNPs) (subsequently referred to as mRNA-LNPs). The primary hypotheses are:

1. the CH505M5 N197D mRNA-gp160 will expand CH235-like B cell precursors,
2. the CH505 TF mRNA-gp160 will boost CH235-like bnAb B cell precursors to acquire more functional mutations needed for broadly neutralizing antibody (bnAb) development, and
3. these mRNA-LNPs will be safe and well tolerated among individuals living without HIV.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrates an understanding of the study and is able and willing to complete the informed consent process.
2. 18 to 55 years old, inclusive, on day of enrollment.
3. Available for clinic follow-up through the last clinic visit and willing to undergo FNA of an axillary lymph node and undergo leukapheresis.
4. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 312 Protocol Safety Review Team (PSRT) are required prior to enrollment into HVTN 312.
5. In good general health according to the clinical judgment of the site investigator.
6. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
7. For US sites: Agrees to discuss their potential for HIV acquisition and agrees to prevention counseling.
8. For non-US sites: Assessed by clinical staff as having a low likelihood of acquiring HIV per guidelines, agrees to discuss their potential for HIV acquisition, agrees to prevention counseling, and agrees to avoid behaviors associated with a higher likelihood of acquiring HIV through the final study visit. "Low likelihood" may include persons stably taking pre-exposure prophylaxis (PrEP) as prescribed.
9. Hemoglobin (Hgb):

   * ≥ 11.0 g/dL for AFAB volunteers
   * ≥ 13.0 g/dL for cisgender AMAB volunteers or for volunteers who have been on masculinizing hormone therapy for more than 6 consecutive months
   * ≥ 12.0 g/dL for AMAB volunteers who have been on feminizing hormone therapy for more than 6 consecutive months
   * For volunteers who have been on gender-affirming hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth.
10. White blood cell (WBC) count = 2,500 to 12,000/mm3 (WBC over 12,000/mm3 is not exclusionary if further evaluation shows general good health and if PSRT approval is granted).
11. Platelets = 125,000 to 550,000/mm3.
12. Alanine aminotransferase (ALT) < 2.5 x upper limit of institutional reference range.
13. Serum creatinine ≤ 1.1 x upper limit of normal (ULN) based on the institutional normal range.
14. Total measured or corrected serum calcium level of > 8.5 mg/dL. Corrected serum calcium should only be used if the total serum calcium is below the lower limit of normal.
15. Systolic blood pressure of 90 to < 140 mmHg and diastolic blood pressure of 50 to < 90 mmHg at screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mmHg systolic and 90 mmHg diastolic. A single measurement ≥ 160 systolic mmHg or 100 mmHg diastolic during the current study evaluation is exclusionary.
16. Negative HIV test results by one of the following options:

    For US volunteers:
    * US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA)
    * Chemiluminescent microparticle immunoassay (CMIA)
    * Two negative results on HIV rapid tests (one of which must be FDA-approved CMIA)

    For non-US volunteers:
    * A negative European Conformity (CE)-marked enzyme immunoassay (EIA)
    * A chemiluminescent microparticle immunoassay (CMIA)
    * A negative result on 2 HIV rapid tests (one of these rapid tests must be CE-marked)
17. Negative for anti-Hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
18. Negative for Hepatitis B surface Ag.
19. For AFAB or intersex at birth volunteers who are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"):

    * Must agree to use effective means of contraception from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.
    * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on the day of enrollment.
20. AFAB or intersex at birth volunteers must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

1. Volunteer who is breastfeeding/chestfeeding or pregnant.
2. Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT approval.
3. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
4. Previous or current recipient of an investigational HIV vaccine or HIV mAb (previous placebo/control recipients are not excluded).
5. Receipt of non-HIV investigational vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) Emergency Use Listing (EUL), or if outside the US, by the national Regulatory Authority (RA) authorizing this clinical trial.
6. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as glucocorticoid use, ≥ prednisone 10 mg/day within 3 months prior to enrollment.
7. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
8. Receipt of any of the following within 4 weeks prior to enrollment:

   * Live replicating vaccine
   * Any mRNA-based vaccine with FDA licensure, FDA EUA, or WHO EUL
   * ACAM2000 vaccine > 28 days prior with a vaccination scab still present.
9. Receipt of any vaccine that is not covered in exclusion criterion #8 within 14 days prior to enrollment. Please note this includes replication-incompetent vaccines such as the Jynneos vaccine for the prevention of mpox disease.
10. History of myocarditis and/or pericarditis.
11. Initiation of Ag-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
12. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of more than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
13. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any mRNA vaccine, including Comirnaty® (Pfizer) and Spikevax® (Moderna), or to any drug administered systemically as a polyethylene glycol containing LNP, including doxorubicin (Doxil, Caelyx, ThermoDox), cisplatin (Lipoplatin) and irinotecan (Onivyde).
14. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
15. Urticaria within the last year unless it was caused by a known, definable, and avoidable trigger (ie, urticaria by a known, definable and avoidable trigger would not be exclusionary).
16. History of chronic urticaria or urticaria previously associated with immunization.
17. Bleeding disorder diagnosed by a clinician that would make study procedures a contraindication.
18. History of seizure(s) within the past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
19. Asplenia or functional asplenia.
20. Active duty and reserve US military personnel.
21. Any other chronic or clinically significant condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of the study participant, hinder their ability to participate in the study, or affect their immune responses to study products. Such conditions include but not limited to: clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgement of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
22. Asthma is excluded if the participant has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days per week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium- to high-dose inhaled corticosteroids (> 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
    * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
23. A participant with a history of a potential immune-mediated medical condition (PIMMC), either active or remote. Not exclusionary: 1) Remote history of Bell's palsy (> 2 years ago) not associated with other neurologic symptoms and 2) mild psoriasis or other mild, uncomplicated, localized or dermatologic condition that does not require ongoing systemic treatment.
24. History of allergy to local anesthetic (Novocain, Lidocaine).
25. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of IV drug use or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of local reactogenicity signs and symptoms after receipt of any study vaccine | Day 15, 71, 127 and 183 (14 days following receipt of any study vaccine)
Frequency of systemic reactogenicity signs and symptoms after receipt of any study vaccine | Day 15, 71, 127 and 183 (14 days following receipt of any study vaccine)
Number of serious adverse events (SAEs) leading to early participant withdrawal or permanent discontinuation | 20 months
Number of medically attended adverse events (MAAEs) leading to early participant withdrawal or permanent discontinuation | 20 months
Number of adverse events of special interest (AESIs) leading to early participant withdrawal or permanent discontinuation | 20 months
Number of adverse events (AEs) leading to early participant withdrawal or permanent discontinuation | 20 months
Response rate of CD4-bs and CH505M5-specific IgG+ B cells as assessed by flow cytometry | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Response rate of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains, as measured by TZM-bl assay | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Magnitude of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains, as measured by TZM-bl assay | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Response rate of differential serum antibody neutralization of precursor detection virus and corresponding epitope KO virus, as measured by the TZM-bl assay | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Magnitude of differential serum antibody neutralization of precursor detection virus and corresponding epitope KO virus, as measured by the TZM-bl assay | Day 127 and 183 (2 weeks after the third and fourth vaccinations)

SECONDARY OUTCOMES:
Response rate of serum IgG binding antibodies to autologous and heterologous HIV Env stabilized trimers, as assessed by binding antibody multiplex assay (BAMA) | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Magnitude of serum IgG binding antibodies to autologous and heterologous HIV Env stabilized trimers, as assessed by BAMA | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Response rate of serum Ab neutralization of heterologous HIV-1 strains as measured by TZM-bl assay | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Magnitude of serum Ab neutralization of heterologous HIV-1 strains as measured by TZM-bl assay | Day 127 and 183 (2 weeks after the third and fourth vaccinations)
Frequency of CD4-bs specific sequences, as measured by BCR single cell sequencing of CD4-bs and CH505M5-specific IgG+ B cells | 20 months
Epitope specific response rates as measured by electron microscopy-based polyclonal epitope mapping (EMPEM) | Day 183 (2 weeks after the fourth vaccination)
Response rate of serum IgG binding Abs to Env Trimers and neutralizing epitopes as assessed by BAMA | Day 337 (24 weeks after the fourth vaccination)
Magnitude of serum IgG binding Abs to Env Trimers and neutralizing epitopes as assessed by BAMA | Day 337 (24 weeks after the fourth vaccination)
Response rate of serum Ab neutralization of autologous, heterologous and precursor HIV-1 strains as measured by TZM-bl assay | Day 337 (24 weeks after the fourth vaccination)
Magnitude of serum Ab neutralization of autologous, heterologous and precursor HIV-1 strains as measured by TZM-bl assay | Day 337 (24 weeks after the fourth vaccination)
Response rate of CD4-bs and CH505M5-specific IgG+ B cells as measured by flow cytometry | Day 337 (24 weeks after the fourth vaccination)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Beth Israel Deaconess Medical Center (Site ID: 32077), Boston, Massachusetts
  - Columbia P&S (Site ID: 30329), New York, New York
  - New York Blood Center (Site ID: 31801), New York, New York
  - Penn Prevention (Site ID: 30310), Philadelphia, Pennsylvania
  - University of Pittsburgh (Site ID: 1001), Pittsburgh, Pennsylvania
  - Seattle Vaccine and Prevention (Site ID: 30331), Seattle, Washington
- Vaccine Trial Centre, Mahidol University CRS (Site ID: 32021), Bangkok, Ratchathewi, Thailand

IPD SHARING:
Plan to Share IPD: No